CLINICAL TRIAL: NCT06744777
Title: The Comparative Efficacy of Standard Treatment Plus Ribavirin vs Standard Treatment Alone in Preventing Clinically Significant Hemorrhage in Patients With Dengue Fever: A Double-blind, Randomized Control Trial
Brief Title: The Comparative Efficacy of Standard Treatment Plus Ribavirin vs Standard Treatment Alone in Preventing Clinically Significant Hemorrhage in Patients With Dengue Fever
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/012
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Severe Dengue
Keywords: Dengue; Hemorrhage; Randomized Controlled Trial; Antiviral Therapy
MeSH Terms: conditions — Dengue; Severe Dengue; Hemorrhage | interventions — Ribavirin

STUDY DESIGN:
Intervention Model Description: The study employs a parallel group design, where participants are randomly assigned to one of two arms: an intervention group receiving standard treatment plus Ribavirin and a control group receiving standard treatment alone. This approach ensures that each participant is exposed to only one of the two interventions being compared. The study is designed to assess the comparative efficacy of Ribavirin in preventing clinically significant hemorrhage among dengue fever patients while minimizing confounding factors through randomization and blinding.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind methodology, with randomization and treatment assignment concealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ribavirin + Standard Treatment (Experimental): Participants in this group will receive the standard treatment for dengue fever alongside Ribavirin. Ribavirin will be administered orally at a dose of 15 mg/kg body weight twice daily (BD) for a total duration of 7 days.
  Interventions: Drug: Ribavirin; Other: Standard Treatment
- Standard Treatment Alone (Active Comparator): Participants in this group will receive only the standard treatment for dengue fever, which includes supportive care such as intravenous fluids and platelet transfusions, as required. No additional pharmacological intervention will be provided.
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Drug: Ribavirin — Ribavirin is an antiviral medication administered as part of the intervention arm. It will be provided orally in a dosage of 15 mg/kg body weight twice daily (BD) for a duration of 7 days. The drug has demonstrated efficacy in vitro and in vivo against RNA viruses, including dengue, through mechanisms such as inosine monophosphate inhibition and immunomodulation.
  Arms: Ribavirin + Standard Treatment
Other: Standard Treatment — The standard treatment for dengue fever includes supportive care measures aimed at managing symptoms and preventing complications. These measures typically involve:
  Intravenous (IV) fluid therapy for rehydration and maintaining hemodynamic stability.
  Platelet transfusion as needed, based on clinical assessment and platelet counts.
  Antipyretics for fever management (excluding non-steroidal anti-inflammatory drugs to prevent bleeding risks).
  Continuous monitoring of vital signs and blood parameters, including platelet counts and hematocrit levels.
  No antiviral drugs or additional pharmacological interventions are included in the standard treatment protocol.

SUMMARY:
This study investigates the comparative efficacy of standard treatment plus Ribavirin versus standard treatment alone in preventing clinically significant hemorrhage among patients diagnosed with dengue fever. It is a double-blind, randomized control trial aimed at determining whether the addition of Ribavirin improves clinical outcomes, particularly reducing bleeding events.

DETAILED DESCRIPTION:
Dengue fever, a significant public health concern, presents varying severity from asymptomatic to life-threatening complications such as hemorrhage or shock. This study evaluates the effectiveness of Ribavirin when combined with standard treatment in mitigating severe bleeding complications in dengue patients. Conducted at multiple public sector hospitals in Khyber Pakhtunkhwa, the trial employs a rigorous methodology, including block randomization, double-blinding, and predefined eligibility criteria. Outcomes include changes in bleeding grades, platelet counts, acute-phase reactants, and hospital stay length. The findings aim to inform policy decisions and enhance dengue fever management protocols.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years and above.
* Hospitalized patients diagnosed with dengue fever, confirmed via:
* Positive Dengue NS1 antigen test
* Dengue IgM antibodies
* Dengue RNA PCR.
* Patients presenting with various severities of illness, as classified by the WHO dengue severity classification.

Exclusion Criteria:

* Patients taking antiplatelet or anticoagulant medications.
* Patients with known bleeding disorders (e.g., hemophilia, von Willebrand disease, end-stage renal disease, or liver cirrhosis).
* Patients with HIV undergoing antiviral therapy.
* Pregnant women.
* Patients with hypersensitivity to Ribavirin.
* Patients with WHO Grade 1 bleeding (few petechiae without clinical significance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Prevention of Clinically Significant Hemorrhage | Up to 7 days post-treatment initiation
  Evaluate the efficacy of Ribavirin plus standard treatment compared to standard treatment alone in preventing clinically significant hemorrhage (WHO Grade 2 or higher).

SECONDARY OUTCOMES:
Platelet Count Changes | At baseline, Day 4, and Day 7 post-treatment initiation.
  Compare levels of platelets count between the intervention and control groups.
Length of Hospital Stay | From hospital admission to discharge (up to 14 days).
  Evaluate and compare the duration of hospitalization in the intervention and control groups.
C-reactive protein | At baseline, Day 4, and Day 7 post-treatment initiation.
  Compare the C-reactive protein in between intervention and control group
Serum ferritin | At baseline, Day 4, and Day 7 post-treatment initiation.
  Compare the serum ferritin in between intervention and control group
Lactate dehydrogenase | At baseline, Day 4, and Day 7 post-treatment initiation.
  Compare levels of lactate dehydrogenase between the intervention and control groups.

OTHER OUTCOMES:
Adverse Events and Tolerability of Ribavirin | During the 7-day treatment period and up to 30 days post-treatment follow-up.
  Document adverse events, including side effects, and assess the tolerability of Ribavirin in the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Said Amin, MBBS,FCPS, Principal Investigator — Department of Medicine Hayatabad Medical Complex Peshawar; Sheraz Fazid, MBBS,MPH, Principal Investigator — Institute of Public Health and Social Science, Khyber Medical University Peshawar; Noman Arif, MBBS, Principal Investigator — Institute of Public Health and Social Science, Khyber Medical University Peshawar; Akhtar Sherin, MBBS,MHR,PHD, Principal Investigator — Kohat Institute of Medical Science Peshawar Pakistan
Locations (4):
- Pakistan (4):
  - Lady Reading Hospital, Peshawar, Khyber Pakhtunkhwa
  - Gandhara Medical Hospital, Peshawar, Khyber Pakhtunkhwa
  - Medical Complex Swabi, Swābi, Khyber Pakhtunkhwa
  - Kohat Institute of Medical Science, Kohat, KPK

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IPD) will be made available to other researchers upon request. This includes data related to demographic information, baseline clinical characteristics, treatment interventions, and outcome measures. Personal identifiers will be removed to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available 6 months after the publication of primary results and remain accessible for 5 years.
Access Criteria: Requests for data sharing will be reviewed by the principal investigator and the ethics committee. Researchers must submit a formal application with a detailed study proposal, including objectives, methodology, and the intended use of the data. A data-sharing agreement will be required to ensure ethical use and data protection compliance.

REFERENCES:
- [Background] Gutierrez E, Sanchez I, Diaz O, Valles A, Balderrama R, Fuentes J, Lara B, Olimon C, Ruiz V, Rodriguez J, Bayardo LH, Chan M, Villafuerte CJ, Padayachee J, Sun A. Current Evidence for Stereotactic Body Radiotherapy in Lung Metastases. Curr Oncol. 2021 Jul 15;28(4):2560-2578. doi: 10.3390/curroncol28040233. PMID 34287274
- [Background] Roy SK, Bhattacharjee S. Dengue virus: epidemiology, biology, and disease aetiology. Can J Microbiol. 2021 Oct;67(10):687-702. doi: 10.1139/cjm-2020-0572. Epub 2021 Sep 3. PMID 34171205
- [Background] Sharif N, Sharif N, Khan A, Dey SK. The Epidemiologic and Clinical Characteristics of the 2023 Dengue Outbreak in Bangladesh. Open Forum Infect Dis. 2024 Feb 2;11(2):ofae066. doi: 10.1093/ofid/ofae066. eCollection 2024 Feb. PMID 38390460
- [Background] Khan U, Azeem S. The rising toll of dengue cases in Pakistan every year: An incipient crisis. Ann Med Surg (Lond). 2022 Mar 31;76:103549. doi: 10.1016/j.amsu.2022.103549. eCollection 2022 Apr. No abstract available. PMID 35495398
- [Background] Gurugama P, Garg P, Perera J, Wijewickrama A, Seneviratne SL. Dengue viral infections. Indian J Dermatol. 2010;55(1):68-78. doi: 10.4103/0019-5154.60357. PMID 20418983
- [Background] Tewari K, Tewari VV, Mehta R. Clinical and Hematological Profile of Patients with Dengue Fever at a Tertiary Care Hospital - An Observational Study. Mediterr J Hematol Infect Dis. 2018 Mar 1;10(1):e2018021. doi: 10.4084/MJHID.2018.021. eCollection 2018. PMID 29531658
- [Background] Ajlan BA, Alafif MM, Alawi MM, Akbar NA, Aldigs EK, Madani TA. Assessment of the new World Health Organization's dengue classification for predicting severity of illness and level of healthcare required. PLoS Negl Trop Dis. 2019 Aug 20;13(8):e0007144. doi: 10.1371/journal.pntd.0007144. eCollection 2019 Aug. PMID 31430283